CLINICAL TRIAL: NCT03865108
Title: Quantifying the Mechanical Environment of Pregnancy Complicated With a Short Cervix With Ultrasound Imaging and Aspiration - Ancillary Study to the Trial of Pessary in Singleton Pregnancies Trial
Brief Title: Mechanical Environment Pregnancy With Short Cervix
Acronym: ATOPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Kristin Myers, Associate Professor of Mechanical Engineering, Columbia University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: AAAO4956 sub-study; 3UG1HD040485-18S1 (NIH)
Record Dates: First submitted 2019-02-22; First posted 2019-03-06 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2024-09

CONDITIONS: Preterm Birth
Keywords: Pessary; Cervix; Biomechanical environment; Aspiration; Computer simulation models
MeSH Terms: conditions — Premature Birth | interventions — High-Energy Shock Waves

STUDY DESIGN:
Intervention Model Description: The two arms are not randomized under this sub study but carried over from the existing TOPS trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pessary and Progesterone (Experimental): Women already receiving a pessary in addition to the standard progesterone through the TOPS trial will undergo ultrasound imaging and cervical speculum examination for information collection.
  Interventions: Procedure: Ultrasound imaging; Procedure: Cervical speculum examination
- Progesterone only (Placebo Comparator): Women already receiving the standard progesterone only will undergo ultrasound imaging and cervical speculum examination for information collection.
  Interventions: Procedure: Ultrasound imaging; Procedure: Cervical speculum examination

INTERVENTIONS:
Procedure: Ultrasound imaging — This standard of care procedure is being done for research purposes and used to collect information and measure the maternal and fetal anatomy.
  Other Names: Sonography
Procedure: Cervical speculum examination — This standard of care procedure is being done for research purposes and used to collect tissue and measure the strength and stiffness of cervix.
  Other Names: Cervical aspiration

SUMMARY:
The objective of this study is to quantify the mechanical environment of pregnancies complicated by a short cervix and randomized in the Trial of Pessary in Singleton Pregnancies with a Short Cervix study with ultrasound imaging and aspiration.

Aim 1: To determine the biomechanical properties of a prematurely remodeled cervix.

Aim 2: To determine the impact of pessary placement on the biomechanical properties of a prematurely remodeled cervix and establish if the pessary reduces the mechanical load on the cervix through computer modeling informed by ultrasonographic measurement and cervical stiffness measurements.

Aim 3: To determine if the differences in the cervical biomechanical properties after pessary placement lead to improved birth outcomes as compared to the progesterone only group.

DETAILED DESCRIPTION:
In pregnancy the mother carries the growing fetus throughout gestation as her body prepares for delivery. This maternal preparation includes anatomical, physiological, and biochemical changes of the uterus, cervix, and ligaments that surround and support the uterus and cervix. For a successful term delivery, the uterus, cervix and supporting ligaments must remodel in a coordinated fashion to allow for adequate dilation and effacement of the cervix and delivery of the fetus.

Preterm birth (PTB) is the leading cause of neonatal death. Premature babies that survive face a significantly increased risk of long-term disabilities, such as mental retardation, learning and behavioral problems, cerebral palsy, seizures, respiratory problems, gastrointestinal problems and vision/hearing loss. PTB is also significant cost factor in healthcare. In 2003, a study in the US approximated neonatal costs to be $224,400 for a newborn that weighed 500-700g (extreme-severe preterm range) verse $1,000 at over 3,000g. These costs increase exponentially with decreasing gestational age and weight. In 2007, an Institute of Medicine report entitled "Preterm Birth" found that the 550,000 preemies born each year in the U.S. cost $26 billion annually, mostly related to prolonged care in neonatal intensive care units. The pathophysiology of PTB is multi-factorial and the degree of severity spans a wide range, with pregnancy outcomes depending on a combination of congenital, anatomical, obstetric, epidemiological, and biochemical factors. Because of these confounding factors PTB rates in the US and around the world are on the rise and diagnostic methods to identify high-risk women for PTB remain elusive.

Premature cervical remodeling which leads to softening/shortening of the cervix (i.e., a mechanical failure of the cervix) is one of the leading contributors to the birth of a severely preterm neonate. The true frequency and impact is unknown because diagnosing this condition remains elusive and the biomechanical environment of pregnancy is unknown. The pathophysiology is hypothesized to be multi-factorial leading to a common feature of a structurally weak and excessively soft cervix that is unable to remain closed and to support the fetus. Recently, it has been demonstrated that these preterm cervical changes may in some cause premature cervical shortening as measured by transvaginal ultrasound imaging. When this occurs, treatment with progesterone suppositories has been demonstrated to reduce the risk of preterm delivery. However, this treatment is not effective in many cases; probably because a short cervix is a late manifestation of the underlying biostructural alterations in the uterus, cervix and supporting ligaments.

Many clinically-relevant advances in the field of orthopedics and gynecology (i.e., assessing the causes of uterine prolapse have been attributed to the accurate biomechanical modeling of the anatomy and tissue properties using finite element analysis (FEA). FEA is a computer simulation that computes tissue stretch (i.e., tissue strain), tissue stress, and reaction forces when external mechanical forces are applied to the system given the tissue's geometric shape and mechanical properties. Lastly, directly measuring the mechanical stiffness of the uterine cervix through use of a simple aspiration device has shown that in normal pregnancy cervical tissue softens starting in the 1st trimester and continues until dilation. These studies have also shown that using a simple mechanical aspirator applied to the end of the cervix protruding into the vaginal canal has zero adverse effects on the patient, where the measurement can be performed during a standard speculum exam.

The cervical pessary has been proposed as an additional option for treatment in pregnancies with a short cervix. It offers additional theoretical benefits over the cerclage, in that it does not require surgical intervention. Its proposed mechanisms of action include a) angling the cervix toward the posterior, bringing the external os toward the sacrum, b) mechanically closing the cervix with the constraining geometry of the device, and c) preserving the mucous plug. These mechanisms of action involve lowering the mechanical stresses on the area of the internal os, potentially modifying the release of the enzymes and inflammatory markers involved in the preterm birth pathway. However, it is still unknown if the pessary relieves the mechanical load on the cervix because a biomechanical investigation of its function has not been performed. Therefore, the investigator plans to study a group of women with a short cervix randomized in an existing trial: AAAR1353 - A Randomized Trial of Pessary in Singleton Pregnancies with a Short Cervix (TOPS) in order to better understand the function and effect of the cervical pessary on the biomechanical support of the cervix in addition to its effect on its tissue properties and structural integrity. If a specific maternal utero-cervical phenotype can be located, where the placement of the cervical pessary reduces the mechanical load on the cervical internal os and therefore leads to a decreased incidence of preterm birth, then a more personalized treatment may be possible for patients who fall within this specific phenotype in the future.

For the substudy, a total of 36 women will be recruited and randomized through the existing TOPS trial (18 randomized to Pessary and Progesterone and 18 randomized to progesterone only). Obstetric and gynecologic history, age, race, body mass index, smoking history, and outcome of the current pregnancy will be recorded for all patients.

ELIGIBILITY:
Inclusion Criteria:

* Singleton gestation.

  * Twin gestation reduced to singleton either spontaneously or therapeutically, is not eligible unless the reduction occurred before 13 weeks 6 days project gestational age.
  * Higher order multifetal gestations reduced to singletons are not eligible.
* Gestational age at randomization between 16 weeks 0 days and 23 weeks 6 days based on clinical information and evaluation of the earliest ultrasound as described in Gestational Age.
* Cervical length on transvaginal examination of less than or equal to 20 mm within 10 days prior to randomization by a study certified sonographer. There is no lower cervical length threshold.

Exclusion Criteria:

* Women who are ineligible for the TOPS trial.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2017-06-05 (Actual); Primary Completion 2021-01-23 (Actual); Study Completion 2021-01-23 (Actual)

PRIMARY OUTCOMES:
Mechanical compliance index of the cervix | Baseline (at diagnosis of short cervix), third trimester (approximately 26-30 weeks)
  The mechanical compliance index of the cervix is the percentage of the cervical tissue above a 1.2 stretch threshold under a uniform IUP. This index is calculated using finite element computational methods, given the maternal anatomy and cervical stiffness measured from the aspiration tool. The mechanical compliance index of the cervix will be measured at both time points within the study timeframe, and the change of the mechanical compliance index between the two time points will be assessed. The main outcome parameter will be the mechanical compliance index at the baseline time point, and the other two outcome measures will be used as validation data points.

SECONDARY OUTCOMES:
Number of participants with spontaneous preterm birth | Pregnancy duration, an average of up to 40 weeks
  The investigator will tally the number of women who receive Intervention of Pessary and experience spontaneous preterm birth

CONTACTS AND LOCATIONS:
Overall Officials: Kristin Myers, PhD, Principal Investigator — Associate Professor of Mechanical Engineering
Locations (1):
- Columbia University Irving Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Lorenz JM. The outcome of extreme prematurity. Semin Perinatol. 2001 Oct;25(5):348-59. doi: 10.1053/sper.2001.27164. PMID 11707021
- [Background] Goldenberg RL, Culhane JF, Iams JD, Romero R. Epidemiology and causes of preterm birth. Lancet. 2008 Jan 5;371(9606):75-84. doi: 10.1016/S0140-6736(08)60074-4. PMID 18177778
- [Background] Gilbert WM, Nesbitt TS, Danielsen B. The cost of prematurity: quantification by gestational age and birth weight. Obstet Gynecol. 2003 Sep;102(3):488-92. doi: 10.1016/s0029-7844(03)00617-3. PMID 12962929
- [Background] Iams JD, Johnson FF, Sonek J, Sachs L, Gebauer C, Samuels P. Cervical competence as a continuum: a study of ultrasonographic cervical length and obstetric performance. Am J Obstet Gynecol. 1995 Apr;172(4 Pt 1):1097-103; discussion 1104-6. doi: 10.1016/0002-9378(95)91469-2. PMID 7726247
- [Background] Beck S, Wojdyla D, Say L, Betran AP, Merialdi M, Requejo JH, Rubens C, Menon R, Van Look PF. The worldwide incidence of preterm birth: a systematic review of maternal mortality and morbidity. Bull World Health Organ. 2010 Jan;88(1):31-8. doi: 10.2471/BLT.08.062554. Epub 2009 Sep 25. PMID 20428351
- [Background] Schmidt H, Galbusera F, Rohlmann A, Shirazi-Adl A. What have we learned from finite element model studies of lumbar intervertebral discs in the past four decades? J Biomech. 2013 Sep 27;46(14):2342-55. doi: 10.1016/j.jbiomech.2013.07.014. Epub 2013 Aug 3. PMID 23962527
- [Background] Ashton-Miller JA, Delancey JO. On the biomechanics of vaginal birth and common sequelae. Annu Rev Biomed Eng. 2009;11:163-76. doi: 10.1146/annurev-bioeng-061008-124823. PMID 19591614
- [Background] Mazza E, Nava A, Bauer M, Winter R, Bajka M, Holzapfel GA. Mechanical properties of the human uterine cervix: an in vivo study. Med Image Anal. 2006 Apr;10(2):125-36. doi: 10.1016/j.media.2005.06.001. Epub 2005 Sep 6. PMID 16143559
- [Background] Bauer M, Mazza E, Nava A, Zeck W, Eder M, Bajka M, Cacho F, Lang U, Holzapfel GA. In vivo characterization of the mechanics of human uterine cervices. Ann N Y Acad Sci. 2007 Apr;1101:186-202. doi: 10.1196/annals.1389.004. Epub 2007 Mar 15. PMID 17363446
- [Background] Mazza E, Nava A, Hahnloser D, Jochum W, Bajka M. The mechanical response of human liver and its relation to histology: an in vivo study. Med Image Anal. 2007 Dec;11(6):663-72. doi: 10.1016/j.media.2007.06.010. Epub 2007 Jul 5. PMID 17719834
- [Background] Bauer M, Mazza E, Jabareen M, Sultan L, Bajka M, Lang U, Zimmermann R, Holzapfel GA. Assessment of the in vivo biomechanical properties of the human uterine cervix in pregnancy using the aspiration test: a feasibility study. Eur J Obstet Gynecol Reprod Biol. 2009 May;144 Suppl 1:S77-81. doi: 10.1016/j.ejogrb.2009.02.025. Epub 2009 Mar 13. PMID 19285777
- [Background] Badir S, Mazza E, Zimmermann R, Bajka M. Cervical softening occurs early in pregnancy: characterization of cervical stiffness in 100 healthy women using the aspiration technique. Prenat Diagn. 2013 Aug;33(8):737-41. doi: 10.1002/pd.4116. Epub 2013 Apr 29. PMID 23553612
- [Background] Badir S, Bajka M, Mazza E. A novel procedure for the mechanical characterization of the uterine cervix during pregnancy. J Mech Behav Biomed Mater. 2013 Nov;27:143-53. doi: 10.1016/j.jmbbm.2012.11.020. Epub 2012 Dec 11. PMID 23274486
- [Background] Hollenstein M, Bugnard G, Joos R, Kropf S, Villiger P, Mazza E. Towards laparoscopic tissue aspiration. Med Image Anal. 2013 Dec;17(8):1037-45. doi: 10.1016/j.media.2013.06.001. Epub 2013 Jun 19. PMID 23876854
- [Background] Mazza E, Parra-Saavedra M, Bajka M, Gratacos E, Nicolaides K, Deprest J. In vivo assessment of the biomechanical properties of the uterine cervix in pregnancy. Prenat Diagn. 2014 Jan;34(1):33-41. doi: 10.1002/pd.4260. PMID 24155152
- [Background] Ginsberg Y, Goldstein I, Lowenstein L, Weiner Z. Measurements of the lower uterine segment during gestation. J Clin Ultrasound. 2013 May;41(4):214-7. doi: 10.1002/jcu.22023. Epub 2013 Mar 16. PMID 23505018
- [Background] Sokolowski P, Saison F, Giles W, McGrath S, Smith D, Smith J, Smith R. Human uterine wall tension trajectories and the onset of parturition. PLoS One. 2010 Jun 23;5(6):e11037. doi: 10.1371/journal.pone.0011037. PMID 20585649
- [Background] Durnwald CP, Mercer BM. Myometrial thickness according to uterine site, gestational age and prior cesarean delivery. J Matern Fetal Neonatal Med. 2008 Apr;21(4):247-50. doi: 10.1080/14767050801926709. PMID 18330820
- [Background] Buhimschi CS, Buhimschi IA, Norwitz ER, Sfakianaki AK, Hamar B, Copel JA, Saade GR, Weiner CP. Sonographic myometrial thickness predicts the latency interval of women with preterm premature rupture of the membranes and oligohydramnios. Am J Obstet Gynecol. 2005 Sep;193(3 Pt 1):762-70. doi: 10.1016/j.ajog.2005.01.053. PMID 16150272
- [Background] Buhimschi CS, Buhimschi IA, Malinow AM, Weiner CP. Myometrial thickness during human labor and immediately post partum. Am J Obstet Gynecol. 2003 Feb;188(2):553-9. doi: 10.1067/mob.2003.77. PMID 12592271
- [Background] Deyer TW, Ashton-Miller JA, Van Baren PM, Pearlman MD. Myometrial contractile strain at uteroplacental separation during parturition. Am J Obstet Gynecol. 2000 Jul;183(1):156-9. doi: 10.1067/mob.2000.105819. PMID 10920324
- [Background] Degani S, Leibovitz Z, Shapiro I, Gonen R, Ohel G. Myometrial thickness in pregnancy: longitudinal sonographic study. J Ultrasound Med. 1998 Oct;17(10):661-5. doi: 10.7863/jum.1998.17.10.661. PMID 9771611
- [Background] Wachsberg RH, Kurtz AB, Levine CD, Solomon P, Wapner RJ. Real-time ultrasonographic analysis of the normal postpartum uterus: technique, variability, and measurements. J Ultrasound Med. 1994 Mar;13(3):215-21. doi: 10.7863/jum.1994.13.3.215. PMID 7932980